CLINICAL TRIAL: NCT04238455
Title: Addition of Ultrasound-Guided Serratus Anterior Plane Block to an Enhanced Recovery Pathway for Thoracoscopic Lung Resection: A Randomized Trial
Brief Title: Ultrasound-Guided Serratus Anterior Plane Block for Additional Pain Relief After Lung Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 19-470
Record Dates: First submitted 2020-01-22; First posted 2020-01-23 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Thoracic Surgery
Keywords: Serratus Anterior Plane Block; segmentectomy; lobectomy; 19-470

STUDY DESIGN:
Intervention Model Description: This is a two-arm randomized study of chest wall nerve blocks for postoperative analgesia after elective minimally invasive lung resection. The two study groups are: (1) usual care plus serratus anterior plane block (treatment arm), and (2) usual care plus sham serratus anterior plane block (control arm).
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Sham Comparator): Sham serratus anterior plane block plus usual car
  Interventions: Procedure: Sham serratus anterior plane block
- Treatment Group (Active Comparator): Serratus anterior plane block plus usual care
  Interventions: Procedure: Serratus anterior plane block

INTERVENTIONS:
Procedure: Sham serratus anterior plane block — The serratus anterior plane block will be performed by the anesthesiology team just prior to emergence from general anesthesia.
  Arms: Control Group
Procedure: Serratus anterior plane block — The serratus anterior plane block will be performed by the anesthesiology team just prior to emergence from general anesthesia.
  Arms: Treatment Group

SUMMARY:
The purpose of this study is to see if an anesthesia technique called serratus anterior plane block may provide additional pain relief for the chest wall after lung surgery. The study will evaluate the effect the serratus anterior plane block technique has on the need for opioids after surgery,the level of pain during recovery, and other aspects of recovery, like whether the patient has nausea and their ability to breathe deeply. The effects of the serratus anterior plane block will be compared to the effects of an inactive (sham) block.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 years of age who are capable of giving consent. English language proficiency is required.
* Undergoing elective minimally invasive (VATS or RATS) anatomic lung resection (segmentectomy or lobectomy) without an epidural.

Exclusion Criteria:

* Pregnancy (Patients must have a negative pregnancy test within 30 days of the operation)
* History of documented anaphylaxis or contraindication to local anesthetics
* History of ipsilateral thoracic surgery. Ipsilateral thoracic surgery indicates any previous thoracoscopic or open (i.e. via thoracotomy) pleural biopsy, lung resection, esophageal surgery, chest wall resection, or other thoracic surgery within the chest cavity. This does not include image-guided lung biopsy. Note: Mediport placement and other procedures performed by a surgeon/proceduralist NOT within the chest cavity are not excluded. Likewise, patients with a history of ipsilateral breast surgery are also not excluded. The purpose is to exclude patients who may have had injury to the intercostal nerves from previous surgery or who have surgically altered anatomy of the hemithorax.
* Patients undergoing bilateral procedures
* Weight < 50 kg
* Chronic sustained-release opioid use for > 2 weeks duration (in the 30 days prior to surgery)
* Significant cognitive impairment or documented psychological impairment
* American Society of Anesthesiologists (ASA) physical status > 3
* Patients may also be excluded from the study if the block is deemed not technically feasible (this may be determined intraoperatively).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
number of patients requiring opioids | within 24 hours post-operation
  Assessment of this outcome will be performed by abstracting total dosage of opioids administered during this time period from the electronic medical record (EMR). Opioid dosages will be converted to intravenous morphine sulfate equivalent.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Jackson, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (6):
- United States (6):
  - Memorial Sloan Kettering Monmouth (Consent only), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent only ), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (Consent Only), Commack, New York
  - Memorial Sloan Kettering Westchester (Consent only), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Consent only), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm